CLINICAL TRIAL: NCT06813976
Title: PRODIGE 98 : Randomized, Multicenter Phase 3 Trial of Adjuvant Chemotherapy With Modified FOLFIRINOX Versus Capecitabine or Gemcitabine in Patients With Resected Ampullary Adenocarcinoma
Acronym: AMPIRINOX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MANFREDI PHRCK 2023
Record Dates: First submitted 2024-12-24; First posted 2025-02-07 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Ampullary Adenocarcinoma
MeSH Terms: interventions — Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental strategy (Experimental)
  Interventions: Drug: mFOLFORINOX; Other: Quality of life questionnaires: QLQ-C30 and PAN26; Biological: Biological assessment; Diagnostic Test: Paraclinical examinations
- Standard treatments (Active Comparator)
  Interventions: Drug: Capecitabine or gemcitabine; Other: Quality of life questionnaires: QLQ-C30 and PAN26; Biological: Biological assessment; Diagnostic Test: Paraclinical examinations

INTERVENTIONS:
Drug: mFOLFORINOX — mFOLFIRINOX every 2 weeks during 12 cycles (24 weeks):
  * Oxaliplatin 85 mg/m²
  * Irinotecan 150 mg/m²
  * Leucovorin 400 mg/m²
  * Fluorouracil 2400 mg/m² during 46 hours
  Arms: Experimental strategy
Drug: Capecitabine or gemcitabine — investigator's choice:
  * Capecitabine 1250 mg/m² BID, 2 weeks on, 1 week off during 8 cycles (24 weeks) OR
  * Gemcitabine 1000 mg/m² in 30 min; 3 weeks on, 1 week of, during 6 cycles ((24 weeks)
  Arms: Standard treatments
Other: Quality of life questionnaires: QLQ-C30 and PAN26 — Before treatment, during treatment (every 12 weeks in any treatment arm Until disease progression or end of follow-up) and after treatment discontinuation (30 days after the end of treatment)
Biological: Biological assessment — Before each course of treatment and between courses of treatment if necessary
Diagnostic Test: Paraclinical examinations — Every 3 months

SUMMARY:
Ampullary adenocarcinoma (AMPAC) is a rare cancer (0.2% of digestive cancers) affecting the ampulla of Vater. The only curative treatment is surgery, but around 4% of patients recur within 2 years of surgical resection.

The aim of adjuvant chemotherapy is to reduce the risk of disease recurrence, and the only chemotherapies that can be considered standard to date are capecitabine and gemcitabine.

In this trial, an alternative experimental treatment strategy using modified FOLFORINOX (mFOLFORINOX) is proposed. It consists of 3 chemotherapies with complementary actions: 5-fluorouracil, irinotecan and oxaliplatin, combined with folic acid a vitamin that enhances the efficacy of 5-fluorouracil.

This study proposes 2 treatment schemes:

* Group A: mFOLFIRINOX: oxaliplatin, irinotecan, 5-fluorouracil, with folinic acid,
* group B: mono-chemotherapy with capecitabine or gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma on surgical specimen
* Macroscopically complete surgical resection of an ampullary adenocarcinoma (R0 or R1)
* Adenocarcinoma removed within 12 weeks prior to enrollment
* Patients ≥ 18 years of age
* Patient without metastatic disease on CT scan < 4 weeks prior to inclusion
* WHO performance status 0 or 1 (WHO 0 if age >75)
* Normal values of kalemia, magnesemia and calcemiaPatient able to understand and sign the information and informed consent note
* Women of childbearing age and men who are sexually active with women of childbearing age must agree to use highly effective contraception during the trial treatment at least until 6 months after the end of experimental treatment. Women of childbearing potential must use highly effective contraception at least 9 months after the end of treatment with oxaliplatin
* Patient affiliated to a social security scheme for France, or equivalents in European countries
* CA19.9 level < 180 U/L at inclusion (post-operative level)

Exclusion Criteria:

* Neoadjuvant systemic chemotherapy
* pT1N0M0 tumors
* Active infection by HBV, HCV or HIV
* Dihydropyrimidine dehydrogenase deficiency (uracilemia ≥ 16 ng/mL)
* Pre-existing peripheral neuropathy (grade ≥ 2)
* Unresolved or uncontrolled concomitant medical conditions
* Neutrophils < 1500/mm3, platelets < 150 000/mm3, Haemoglobin < 9 g/dL
* Total bilirubin > 1.5x normal,
* Creatinine clearance < 50 ml/min according to MDRD
* AST or ALT > 2.5 x UNL, alkaline phosphatase > 2.5x normal at least 15 days after resection
* Patients with poor nutritional status represented by albuminemia < 30.0g/dl
* History of myocardial infarction within the last 6 months, severe coronary artery disease or severe heart failure
* Active and/or potentially severe infection
* Treatment with a strong cytochrome P450 inhibitor within 4 weeks prior to the administration of the protocol treatment (Treatment with Hypericum perforatum)
* Patient under treatment by brivudine, or treated by brivudine within 4 weeks prior to beginning of study treatment
* Concomitant use with St John's Wort
* QT/QTc interval longer than 450msec for men and longer than 470msec for women on the ECG
* Hypersensitivity to any of the study products or their excipients
* Administration of live vaccines within 28 days prior to randomization
* Other cancer treated within the last 5 years except adequately treated, in situ cervical carcinoma or basocellular/spinocellular carcinoma
* chronic bowel disease requiring specific treatment and/or intestinal obstruction
* Pregnant or breastfeeding woman
* Person under guardianship
* Inability to undergo the medical follow-up of the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2033-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Assessed up to 36 months
  To compare DFS between the 2 arms of treatments in randomized patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France